CLINICAL TRIAL: NCT04891445
Title: Efficacy of a Nursing Monitoring Program for Detection and Treatment of Hepatitis C in a Population With Severe Mental Disorder.
Brief Title: Hepatitis C in Severe Mental Disorders: Nursing Programme
Acronym: HEPASAME21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Malaga (Other)
Collaborators: University of Malaga (Other); Gilead Sciences (Industry); Instituto de Investigacion Biomedica de Malaga (Other)
Responsible Party: Principal Investigator, Casta Quemada-González, Mental Health Nursing, Hospital Regional de Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CQG-20 (0444-N-20)
Record Dates: First submitted 2021-04-14; First posted 2021-05-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis C; Severe Mental Disorder
Keywords: Clinical Paths; Patient Care Planning; Hepatitis C; Severe Mental Disorders
MeSH Terms: conditions — Hepatitis C; Mental Disorders | interventions — Critical Pathways

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- As usual (Active Comparator): Patients will be directly referred to their family doctor with a report on the data obtained in the analysis (presence of HCV and positive viral load), so that they can follow the usual treatment (as usual) in these cases in the Andalusian Health Service.
  The usual treatment implies, once the presence of Virus C has been confirmed, referral by the patient's family doctor to the specialized service, in this case the Gastroenterology Service of the referral Hospital, through the usual appointment procedure. Generally the delay in this process is usually approx. 2-3 months for the first appointment.
  Interventions: Behavioral: As usual
- Nurse-Navigation Programme (Experimental): A Clinical Pathway (CP) of nursing monitoring will be activated, that is, patients will be accompanied throughout the evaluation and treatment process until their complete cure is guaranteed.
  CP will include the activation of care in the Gastroenterology Service by the nurse. By requesting a first appointment in the Gastroenterology Service, via email, the nurse will activate the patients' access to this first appointment, which consist in a one-step intervention: liver evaluation analysis on the genotype, determine the most appropriate type of treatment and, dispensing treatment by the Hospital Pharmacy Unit. To guarantee attendance, in all cases the patient will be accompanied, either by a competent available family caregiver, or by the mental health nursing team.
  All the intervention will be operationalized through the mentioned CP developed for this purpose, with the participation of those involved.
  Interventions: Behavioral: Nursing monitoring program

INTERVENTIONS:
Behavioral: Nursing monitoring program — A clinical pathway will be activate that allows all the necessary interventions, once the person is diagnosed, to be carried out on the same day, and a mental health nursing team will monitor the entire process.
  Other Names: Clinical Path
  Arms: Nurse-Navigation Programme
Behavioral: As usual — Referral to the family doctor for a request for follow-up by the gastroenterologist. The specialist prescribes the tests for the definitive diagnosis that will take place in other units (with their corresponding appointments). After this, the patient will return to the specialist to establish the treatment to follow. Pharmacological treatment will be dispensed at the hospital pharmacy (collected once a month until completion of treatment and confirmation of cure). This last step of the treatment will be done in a new consultation at the gastroenterology service after blood tests to verify the disappearance of the viral load.
  Arms: As usual

SUMMARY:
It has been described in the scientific literature that people diagnosed with serious mental disorders, such as psychosis and schizophrenia, have difficulties to access medical treatments for their physical illnesses, which produces excess mortality in this population.

This project will consist of three different parts. The first will be the detection and accurate diagnosis of hepatitis C (HCV) in the population diagnosed with a severe mental disorder (SMD). It will find the prevalence of people with infection who have not been diagnosed, as well as that of people diagnosed but who have not completed treatment. Likewise, the characteristics of the sample obtained and the risk factors associated with positive cases will be analyzed.

The second part of the study will consist of comparing the effectiveness of an individualized monitoring programme (NURSE-NAVIGATION PROGRAMME), carried out by the specialist mental health nurse, during the treatment of hepatitis C versus the usual health care.

In order to fulfill these first two objectives, a Clinical Pathway will be opened in which the Microbiology, Gastroenterology, Pharmacy and Mental Health services of the Regional University Hospital of Malaga will participate.

The third objective of the project will be to study how the presence of Hepatitis C influences psychotic symptoms, mainly negative ones, changes in daily functioning and changes in quality of life . For these purposes we will use the PANSS scale, a Quality of Life scale (the Life Skill Profile) and the Euroqol5D Health Questionaire before treatment and after verifying the effective cure of HCV.

A third and final evaluation with all the study variables will be carried out 6 months after starting the treatment. In addition, the disappearance of the viral load and, therefore, the patient's cure will be determined with a new blood test.

DETAILED DESCRIPTION:
The objective of this study is to compare the effectiveness of a nurse-navigation program developed by specialist nurses on mental health, for patients with HCV and SMD, against the usual standard care, regarding the detection of the disease, facilitation of access and adherence to treatment, guides through the healthcare system, and cure from HCV.

The null hypothesis that this study will test is that there are no differences in the HCV cure rate in SMD subjects who receive the nurse-navigation model versus those who receive usual care. Additionally, a second hypothesis will be tested regarding to the differences in the adherence to HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Severe mental disorder
* Hepatitis C positive with viral load

Exclusion Criteria:

* Patients who have contraindicated HCV treatment for any reason
* Patients in a clear situation of psychopathological decompensation (until recovery)
* Patients does not agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Healing | 6 months
  % healing in both groups (measured as undetectable viral load in a blood test done 3 months after finishing treatment).
Adherence | 8-12 weeks
  Adherence to treatment in both groups using AIDS Clinical Trials Group method (medications not taken in a period of 4 days prior to the interview: % adherence = (total galenic units prescribed for that period - total units not taken) / total galenic units prescribed for that period)

SECONDARY OUTCOMES:
Changes in daily functioning | 6 months
  Changes in daily functioning, measured with Life Skill Profile (LSP) where a higher score means better daily functioning.
Negative symptoms | 6 months
  Negative symptoms, measured with Positive and Negative Syndrome Scale PANSS, with 30 items that are scored from 1-absent to extreme 7 symptoms where a higher score indicates greater severity of symptoms
Changes in health related quality of life | 6 months
  Health related quality of life is assessed by the European Quality of Life-5 Dimensions Questionnaire (EQ-5D). A higher score means better health.
Detection rate | 2 years
  % Detection after screening the severe mental disorder population

OTHER OUTCOMES:
Characterization variable 1 | At the beginning
  Age (in years)
Characterization variable 2 | At the beginning
  Sex (male / female)
Characterization variable 3 | At the beginning
  Type of diagnosis (classification according to DSM-IV)
Characterization variable 4 | At the beginning
  Disease evolution time (in months)
Characterization variable 5 | At the beginning and if there are changes (6 months)
  Drug treatment (name and dose of all drugs)
Characterization variable 6 | At the beginning and if there are changes (6 months)
  Physical comorbidities according to the list of physical diseases proposed by Diederichs et al. (2011) (cancer, diabetes mellitus, hypertension, myocardial infarction, chronic ischemic heart disease, cardiac arrhythmias, heart failure, cerebrovascular accident, chronic obstructive pulmonary disease and arthritis).
Characterization variable 7 | At the beginning and if there are new hospital admission (6 months)
  Number of admissions to a mental health hospitalization unit in the last 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: María Magdalena Hurtado, PhD, Study Chair — Regional Hospital of Málaga, Spain.; Celia Martí-García, PhD, Study Chair — Faculty of Health Sciences. University of Málaga, Spain; José Miguel Morales-Asencio, PhD, Study Director — Faculty of Health Sciences. University of Málaga, Spain.; Casta Quemada, Principal Investigator — Regional Hospital of Málaga, Spain.
Locations (1):
- Regional Hospital of Málaga, Málaga, Malaga, Spain

REFERENCES:
- [Derived] Quemada-Gonzalez C, Morales-Asencio JM, Hurtado MM, Marti-Garcia C. Study protocol: a randomised, controlled trial of a nurse navigator program for the management of hepatitis C virus in patients with severe mental disorder. BMC Nurs. 2022 Apr 20;21(1):92. doi: 10.1186/s12912-022-00870-w. PMID 35443727